CLINICAL TRIAL: NCT03490838
Title: A Phase 1/2 Open-label, Multi-center, Dose-escalation Study of Safety, Tolerability, Pharmacokinetics, Dosimetry, and Response to Repeat Dosing of 177Lu-PSMA-R2 Radio-ligand Therapy in Patients With Prostate Specific Membrane Antigen (PSMA) Positive (68Ga-PSMA-R2) Progressive Metastatic Castration-resistant Prostate Cancer, Following Previous Systemic Treatment
Brief Title: 177Lu-PSMA-R2 in Patients With PSMA Positive Progressive, Metastatic, Castration Resistant Prostate Cancer
Acronym: PROter
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment for PROter A206T-G01-001 (NCT03490838) was halted in Phase I by sponsor decision. Phase II expansion portion of the study was never initiated.
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A206T-G01-001; 2017-004034-29 (EudraCT Number); CAAA602A12101 (Other: Novartis)
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasm
Keywords: Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Prostatic Diseases; Cancer of Prostate; Cancer of the Prostate; Neoplasms, Prostate; Neoplasms, Prostatic; Prostate Cancer; Prostate Neoplasms; Prostatic Cancer; Prostate-Specific Membrane Antigen; PSMA; PSMA radioligand therapy
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase I: Dose Escalation Cohort 1 (Experimental): 3.70 GBq (100 mCi) x 3 times
  Interventions: Drug: 177Lu-PSMA-R2
- Phase I: Dose Escalation Cohort 2 (Experimental): 7.40 GBq (200 mCi) up to 4 times
  Interventions: Drug: 177Lu-PSMA-R2
- Phase I: Dose Escalation Cohort 3 (Experimental): 11.1 GBq (300 mCi) up to 4 times
  Interventions: Drug: 177Lu-PSMA-R2
- Phase I: Dose Escalation Cohort 4 (Experimental): 14.8 GBq (400 mCi) up to 4 times
  Interventions: Drug: 177Lu-PSMA-R2
- Phase I: Dose Escalation Cohort 5 (Experimental): 18.5 GBq (500 mCi) up to 4 times
  Interventions: Drug: 177Lu-PSMA-R2
- Phase I: Dose Escalation Cohort 6 (Experimental): 18.5 GBq (500 mCi) up to 3 times
  Interventions: Drug: 177Lu-PSMA-R2

INTERVENTIONS:
Drug: 177Lu-PSMA-R2 — radio-ligand therapy

SUMMARY:
This Phase 1/2 study is intended to investigate the safety, tolerability, and radiation dosimetry of 177Lu-PSMA-R2 and further assess preliminary efficacy data in patients with metastatic castration-resistant prostate cancer (mCRPC). The Phase 1 portion of the study will determine the recommended dose of 177Lu-PSMA-R2 for radio-ligand therapy (RLT) of mCRPC, and the Phase 2 portion will expand into approximately 60 patients documenting the preliminary activity (anti-tumor response) of repeated treatments administered, continuing safety assessments and collecting QoL data.

DETAILED DESCRIPTION:
Recruitment for PROter A206T-G01-001 (NCT03490838) was halted in Phase I by sponsor decision. Phase II expansion portion of the study was never initiated. Importantly, this recruitment halt was not a consequence of any safety concern. Ongoing patients at the time of recruitment halt continued per protocol and completed the 1 year safety follow-up prior to early study termination.

The primary objective of the Phase I portion of the study to assess the safety and tolerability of 177Lu-PSMA-R2 and to assess Dose Limiting Toxicities (DLTs) and determine the maximum tolerated dose (MTD) (if reached) and the recommended Phase II dose was not reached due to early recruitment halt.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, 18 years of age or older
* Signed and dated written ICF by the patient or legally acceptable representative prior to any study-specific procedures
* Histologically confirmed adenocarcinoma of the prostate
* Serum testosterone levels < 50 ng/dL after surgical or continued chemical castration
* Metastatic disease documented by CT/MRI or bone scan (not older than 28 days at enrollment) revealing at least one metastatic lymph-node, visceral metastasis and/or bone metastasis
* Positive 68Ga-PSMA-R2 PET/CT scan for central eligibility assessment. Patients who receive 68Ga-PSMA-R2 as part of separate clinical protocol are eligible (must meet all study eligibility criteria)
* Documented progressive mCRPC on or after the last systemic treatment administered for the advanced disease including metastatic disease. Disease progression defined as increasing serum PSA (per PCWG3), radiological progression or ≥ 2 new bone lesions.
* Must have received prior systemic treatment for mCRPC including CYP17 inhibitors and/or androgen-pathway inhibitors (i.e. abiraterone and/or enzalutamide when available) and one and no more than one line of chemotherapy for the advanced disease (unless ineligible (unfit) to receive chemotherapy).
* At least 28 days elapsed between last anti-cancer treatment administration and the initiation of study treatment (except for Luteinizing Hormone-releasing Hormone [LHRH] or Gonadotropin-releasing Hormone [GnRH]), or resolution of all previous treatment related toxicities to CTCAE version 5.0 grade of ≤ 1 (except for chemotherapy induced alopecia and grade 2 peripheral neuropathy or grade 2 urinary frequency which are allowed). Prior major surgery must be at least 12 weeks prior to study entry.
* Eastern cooperative oncology group (ECOG) performance status of 0-2 with a life expectancy ≥ 6 months
* Adequate bone marrow reserve and organ function as demonstrated by complete blood count, and biochemistry in blood and urine at baseline

  1. Platelet count of >100 x10e9/L
  2. White blood cell (WBC) count > 3,000/mL
  3. Neutrophil count > 1,500/mL
  4. Hemoglobin ≥ 10 g/dL
  5. Serum creatinine < 1.5 x upper limit normal (ULN) or estimated glomerular filtration rate (GFR) > 50 mL/min based upon Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) equation. Patients with estimated GFR between 50 - 60 mL/min at baseline will require a 99mTc-DTPA GFR test and only patients with non-obstructive pathology will be included in the study.
  6. Total bilirubin < 3 x ULN (except if confirmed history of Gilbert's disease)
  7. Baseline serum albumin > 30 g/L
  8. Aspartate aminotransferase (AST) < 3 times the ULN
* For male patients with partners of childbearing potential, agreement to use barrier contraceptive method (condom) and to continue its use for 6 months from receiving the last dose of IP

Exclusion Criteria:

* Pathological finding consistent with small cell, neuroendocrine carcinoma of the prostate or any other histology different than adenocarcinoma.
* Diffuse bone-marrow involvement (i.e. "superscan" defined as bone scintigraphy in which there is excessive skeletal radioisotope uptake [>20 bone lesions] in relation to soft tissues along with absent or faint activity in the genitourinary tract due to diffuse bone/ bone marrow metastases)
* Prior exposure to radioligand therapy radioisotope therapy (e.g. 89Sr), systemic radiotherapy or 223Ra-therapy.
* Current severe urinary incontinence, hydronephrosis, severe voiding dysfunction, any level of urinary obstruction requiring indwelling/condom catheters
* Spinal cord compression or brain metastases
* Uncontrolled pain that results in patient's lack of compliance with the imaging procedures
* Uncontrolled cardiovascular history, defined as:

  * Congestive heart failure (New York Heart Association [NYHA] II, III, IV)
  * Mean resting corrected QT interval (QTc) >450 millisecond (msec), obtained from 3 ECGs recordings, using the screening clinic ECG machine-derived QTc value.
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
  * Any factor increasing the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives, or any concomitant medication known to prolong the QT interval.
* Other known co-existing malignancies except non-melanoma skin cancer or low grade superficial bladder cancer unless definitively treated and proven no evidence of recurrence for 5 years.
* History of deep vein thrombosis and/or pulmonary embolism within 4 weeks of enrollment.
* Known incompatibility to CT or PET scans.
* Any evidence of severe or uncontrolled systemic or psychiatric diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Active infection including human immunodeficiency virus (HIV) and untreated hepatitis B, and hepatitis C. Screening for chronic conditions is not required.
* Patients who have received any investigational treatment agent within the last 28 days.
* Known allergies, hypersensitivity, or intolerance to the IP or its excipients
* Known history of myelodysplastic syndrome/leukemia at any time
* Patient is unlikely to comply with study procedures, restrictions and requirements and judged by the Investigator that the patient is not suitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of dose limiting toxicities (DLTs) during first cycle of study treatment. | Up to 8 weeks after the first 177Lu-PSMA-R2 dose
  A dose-limiting toxicity (DLT) is defined as any toxicity not attributable to the disease or disease-related processes under investigation, the time window for DLT assessment period is Cycle 1. To be considered a DLT, it must be related to the IP (attributions: possible, probable, and definite) while fulfilling one of the following criteria as per the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Phase II: Prostate-Specific Antigen (PSA) response rate 50 | Week 13 (12 weeks after the first 177Lu-PSMA-R2 injection)
  PSA response rate 50 is defined as the proportion of participants who have a greater or equal 50% in PSA from Baseline that is confirmed by a second PSA measurement 4 weeks later, as per Prostate Cancer Working Group 3 (PCWG3) criteria.

SECONDARY OUTCOMES:
Phase I and II: Treatment Emergent Adverse Event (TEAE) rate | From randomization till 30 days safety follow-up, assessed up to 4 years (estimated final OS analysis)
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Phase I and II: Objective Response Rate (ORR) | From date of randomization assessed up to 4 years (estimated final OS analysis)
  ORR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) per RECIST 1.1.
Phase I and II: Duration of Response (DoR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 4 years (estimated final OS analysis)
  Duration of Response (DoR) according to RECIST v1.1 is defined as the time that measurement criteria are met for objective response (CR/PR) (whichever status is recorded first) until the first date of progression or death is documented.
Phase I and II: Prostate-Specific Antigen (PSA) response rate 30 | Week 13 (12 weeks after the first 177Lu-PSMA-R2 injection)
  PSA response rate 30 is defined as the proportion of participants who have a greater or equal 30% in PSA from Baseline that is confirmed by a second PSA measurement 4 weeks later, as per Prostate Cancer Working Group 3 (PCWG3) criteria.
Phase I: Prostate-Specific Antigen (PSA) response rate 50 | Week 13 (12 weeks after the first 177Lu-PSMA-R2 injection)
  PSA response rate 50 is defined as the proportion of participants who have a greater or equal 50% in PSA from Baseline that is confirmed by a second PSA measurement 4 weeks later, as per Prostate Cancer Working Group 3 (PCWG3) criteria.
Phase I: 177Lu-PSMA-R2 plasma concentration | Days 1 through 8 post-treatment
Phase I: Maximum plasma concentration (Cmax) of 177Lu-PSMA-R2 | Day 1 (before the start of infusion, at the mid-point, and just before the end of infusion, then at post infusion at approximately 5, 15, 30 minutes, 1, 2, 4, 6, 8, 24, 40 (+/- 4 hours), 48 hours), Day 4 (+2 days) and Day 8 post end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Phase I: Minimum plasma concentration (Cmin) of 177Lu-PSMA-R2 | Day 1 (before the start of infusion, at the mid-point, and just before the end of infusion, then at post infusion at approximately 5, 15, 30 minutes, 1, 2, 4, 6, 8, 24, 40 (+/- 4 hours), 48 hours), Day 4 (+2 days) and Day 8 post end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmin will be listed and summarized using descriptive statistics.
Phase I: Area under the plasma concentration-time curve (AUC) of 177Lu-PSMA-R2 | Day 1 (before the start of infusion, at the mid-point, and just before the end of infusion, then at post infusion at approximately 5, 15, 30 minutes, 1, 2, 4, 6, 8, 24, 40 (+/- 4 hours), 48 hours), Day 4 (+2 days) and Day 8 post end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC will be listed and summarized using descriptive statistics.
Phase I: Dosimetry | Days 1 through 8 post-treatment
  Radiation (Gy, Gy/MBq) update by critical organs and metastatic lesions
Phase I and II: Patient Reported Outcomes (PRO) of Mouth Dryness using Xerostomia Questionnaire | Prior to dosing on Day 1 and every 12 weeks until 1 year after disease progression or early study termination whichever comes first
  The Xerostomia questionnaire is a questionnaire used to describe mouth dryness and its effects on daily life. It consists of 8 questions with each question score ranging from 0 ("never"/"none") to 10 ("worst"). The sum of the 8 scores produces a total score (score range from 0-80). A low score corresponds to a good quality of life while a high score means a poor quality of life due to the dry mouth.
Phase I and II: Patient Reported Outcomes (PRO) of Eye Dryness using Xerophthalmia Questionnaire | Prior to dosing on Day 1 and every 12 weeks until 1 year after disease progression or early study termination whichever comes first
  The Xerophthalmia questionnaire is a questionnaire used to describe eye dryness and its effects on daily life. It consists of 3 questions. The first 2 questions scores range from 1 ("never") to 4 ("constantly") and the last question is a Yes/No question about previous dry eye diagnosis. The sum of the scores of the first 2 questions produces a total score (score range from 2-8). A low score corresponds to a good quality of life while a high score means a poor quality of life due to the dry eye.
Phase I and II: Brief Pain Inventory-short Form (PBI-SF) | Prior to dosing on Day 1 and every 12 weeks until 1 year after disease progression or early study termination whichever comes first
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item self report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Phase II: Disease Control Rate (DCR) | From date of randomization till 30 days safety fup, assessed up to 4 years (estimated final OS analysis)
  DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST 1.1.
Phase II: Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 4 years (estimated final OS analysis)
  rPFS is defined as the time to radiographic progression by PCWG3-modified RECIST v1.1 or death.
Phase II: Overall Survival (OS) | From date of randomization until date of death from any cause, assessed up to 4 years (estimated final OS analysis)
  OS is defined as the time to death for any cause.
Phase II: Time to Prostate Specific Antigen (PSA) progression | From date of randomization until date of death from any cause, assessed up to 4 years (estimated final OS analysis)
  PSA progression is defined as the time from the date of first dose of 177Lu-PSMA-R2 injection to the first date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained 3 or more weeks later.
Phase II: Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Score | Prior to dosing on Day 1 and every 12 weeks until 1 year after disease progression or early study termination whichever comes first
  The EORTC QLQ-C30 contains 30 questions assessed by the participant. There are 9 multiple-item scales: 5 scales that assess aspects of functioning (physical, role functioning, cognitive, emotional, and social); 3 symptom scales (Fatigue, Pain, and Nausea and Vomiting); and a global health status/Quality of Life (QOL) scale. There are 5 single-item measures assessing additional symptoms (i.e., dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and a single item concerning perceived financial impact of the disease. All but two questions have 4 point scales ranging from "Not at all" to "Very much." The two questions concerning global health status/ QOL have 7 point scales with ratings ranging from "Very poor" to "Excellent." For each of the 14 domains, final scores are transformed such that they range from 0-100, where higher scores indicate improvement.
Phase II: Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Prostate Module (EORTC QLQ-PR25) Score | Prior to dosing on Day 1 and every 12 weeks until 1 year after disease progression or early study termination whichever comes first
  The EORTC QLQ-PR25 is a prostate cancer module for the assessment of health-related quality of life (HRQoL). It consists of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Questions use a 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (9):
  - Pheonix Molecular Imaging Center, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Yale New Haven Children Hospital, New Haven, Connecticut
  - Tulane Cancer Center Tulance Cancer, New Orleans, Louisiana
  - John Hopkins University - Kimmel Comp. Cancer Center, Baltimore, Maryland
  - National Institute of Health, Bethesda, Maryland
  - Mount Sinai Hospital School of Medicine, New York, New York
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center, Madison, Wisconsin
- Spain (2):
  - Hospital Vall Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18023